CLINICAL TRIAL: NCT00293046
Title: A Randomised, Parallel-Group, Open, Controlled Phase III Trial Assessing the Treatment Compliance With GRAZAX® in Subjects With Seasonal Grass Pollen Induced Rhinoconjunctivitis
Brief Title: Assessment of Grazax® Treatment Compliance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GT-10
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Allergy
Keywords: Allergy
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Biological: ALK Grass tablet - use of compliance device

SUMMARY:
This trial is performed to assess whether the Grazax® treatment compliance can be improved by use of a compliance device (Memozax®).

ELIGIBILITY:
Inclusion Criteria:

* Grass pollen induced rhinoconjunctivitis
* Males and females, 18-65 years of age
* Positive skin prick test

Exclusion Criteria:

* Previous treatment with grass pollen allergen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2006-02; Primary Completion 2006-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Assessment of treatment compliance by recording of drug accountability

SECONDARY OUTCOMES:
Recording of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kim Simonsen, MD, Study Director — ALK-Abelló A/S
Locations (1):
- Allgergie - Ambulatorium Rennweg, Vienna, Austria